CLINICAL TRIAL: NCT04331366
Title: GO2 PEEP Study: The Use of a Bidirectional Oxygenation Valve in the Management of Pulmonary Complications of COVID-19
Brief Title: Bidirectional Oxygenation Valve in the Management of Pulmonary Complications of COVID-19
Acronym: GO2 PEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jeffrey Miller, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00000381
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Results first posted 2021-02-10 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
Keywords: Bidirectional oxygenation; Pulmonary compromise; Supplemental oxygen
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment with GO2 PEEP MOUTHPIECE (Experimental): Participants receiving treatment with the GO2 PEEP MOUTHPIECE
  Interventions: Device: GO2 PEEP MOUTHPIECE

INTERVENTIONS:
Device: GO2 PEEP MOUTHPIECE — The GO2 PEEP MOUTHPIECE has a bidirectional valve that delivers PEEP with each breath. Participants will be provided a G02 PEEP MOUTHPIECE to use underneath the oxygen face mask and will be instructed to breathe slowly and deeply through the mouthpiece for 15 minutes total. Metrics for primary and secondary endpoints will be recorded immediately prior to use and then at 5, 10 and 15 minutes of use and then 15 minutes after cessation of use.

SUMMARY:
The objective of this study is to determine the safety, feasibility and efficacy of a bidirectional oxygenation Positive End Expiratory Pressure (PEEP) mouthpiece in coronavirus disease 2019 (COVID-19) patients requiring supplemental oxygen by non-rebreather mask.

DETAILED DESCRIPTION:
Severe cases of COVID-19 often mimic the typical course of Adult Respiratory Distress Syndrome (ARDS) and its predictable sequelae. These patients often require intubation and ventilator support in order to sustain adequate oxygenation. Once a COVID-19 patient is intubated, Positive End Expiratory Pressure (PEEP) is a mainstay of treatment and is used in order to improve lung function, treat underlying atelectasis, improve oxygenation, and improve survival. In fact, early clinical data as well as reports from front line physicians treating COVID-19 suggest that PEEP has been the most effective treatment modality. In many cases, PEEP has resulted in improved oxygenation and improved survival.

PEEP decreases the propensity for the alveoli to collapse by increasing the air pressure in the lungs. This residual pressure in the lungs at the end of exhalation decreases shunting and allows for more complete gas exchange and improved oxygenation. In patients, PEEP is one of the safest ways to increase partial pressure of oxygen (PaO2) and is used on almost all modern ventilator settings.

The GO2 PEEP MOUTHPIECE is a simple, comfortable, and straightforward mouthpiece with a bidirectional valve that effectively delivers PEEP with every breath. Early application of the GO2 PEEP MOUTHPIECE in non-intubated COVID-19 patients may improve outcomes and save lives. Furthermore, this device may allow for less strain on limited resources, especially ventilators. This PEEP mouthpiece could be employed under an oxygen non-rebreather mask to improve oxygenation and avoid intubation.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive
* Oxygen saturation <92%
* Able to provide informed consent
* Receiving oxygen by non-rebreather mask
* Not currently requiring intubation

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Cognitive impairment
* Rapidly decompensating status requiring urgent or emergent higher level of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Emory Saint Joseph's Hospital and Emory University Hospital in Atlanta, Georgia. Enrollment began on April 8, 2020 and all follow up was complete by August 31, 2020.
Groups:
- GO2 PEEP MOUTHPIECE: Participants receiving treatment with the GO2 PEEP MOUTHPIECE.
Period: Overall Study
Arm/Group | GO2 PEEP MOUTHPIECE
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GO2 PEEP MOUTHPIECE
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.71 (21.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation by Pulse Oximetry
Description: Pulse oximetry is a way to assess whether or not a patient needs help breathing. Oxygen saturation levels for healthy individuals are 95% and above.
Time Frame: Baseline, Minutes 5, 10, 15, 30 (15 minutes after treatment ends)
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | GO2 PEEP MOUTHPIECE
Number analyzed (Participants) | 2
percentage of oxygen saturation
  Baseline | 92 (0)
  Minute 5 | 93.5 (0.707)
  Minute 10 | 94 (1.414)
  Minute 15 | 94 (1.414)
  Minute 30 (15 minutes post-treatment) | 92.5 (0.707)

2. Secondary Outcome: Respiratory Rate
Description: The number of breaths per minute was assessed before treatment, during treatment, and 15 minutes after the end of treatment.
Time Frame: Baseline, Minutes 5, 10, 15, 30 (15 minutes after treatment ends)
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | GO2 PEEP MOUTHPIECE
Number analyzed (Participants) | 2
breaths per minute
  Baseline | 23.5 (0.707)
  Minute 5 | 20 (0)
  Minute 10 | 18 (0)
  Minute 15 | 17 (1.414)
  Minute 30 (15 minutes post-treatment) | 18.5 (0.707)

3. Secondary Outcome: Heart Rate
Description: Heart rate, in beats per minute, was assessed before treatment, during treatment, and 15 minutes after the end of treatment.
Time Frame: Baseline, Minutes 5, 10, 15, 30 (15 minutes after treatment ends)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | GO2 PEEP MOUTHPIECE
Number analyzed (Participants) | 2
beats per minute
  Baseline | 84.5 (17.678)
  Minute 5 | 87.5 (17.678)
  Minute 10 | 90.5 (20.506)
  Minute 15 | 86.5 (16.263)
  Minute 30 (15 minutes post-treatment) | 86.5 (14.849)

4. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure was assessed before treatment, during treatment, and 15 minutes after the end of treatment.
Time Frame: Baseline, Minutes 5, 10, 15, 30 (15 minutes after treatment ends)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GO2 PEEP MOUTHPIECE
Number analyzed (Participants) | 2
mmHg
  Baseline Systolic | 152.5 (31.820)
  Baseline Diastolic | 65 (7.071)
  Minute 5 Systolic | 155 (21.213)
  Minute 5 Diastolic | 72.5 (10.607)
  Minute 10 Systolic | 150 (21.213)
  Minute 10 Diastolic | 70 (0)
  Minute 15 Systolic | 145 (21.213)
  Minute 15 Diastolic | 67.5 (3.536)
  Minute 30 (15 minutes post-treatment) Systolic | 152.5 (24.749)
  Minute 30 (15 minutes post-treatment) Diastolic | 65 (7.071)

5. Secondary Outcome: Count of Participants With Subjective Work of Breathing
Description: Participants were observed for stridor, grunting, nasal flaring, or accessory muscle use. The presence of any of these indicates that increased effort is required for breathing.
Time Frame: Baseline, Minutes 5, 10, 15, 30 (15 minutes after treatment ends)
Population: Data on subjective work of breathing were not collected at the Baseline and Minute 30 time points.
Measure: Count of Participants; unit: Participants
Arm/Group | GO2 PEEP MOUTHPIECE
Number analyzed (Participants) | 2
Participants
  Baseline: number analyzed (Participants) | 0
  Minute 5 | 1
  Minute 10 | 0
  Minute 15 | 0
  Minute 30 (15 minutes post-treatment): number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events on the day of the intervention beginning just prior to treatment with the mouthpiece through 15 minutes after the cessation of PEEP therapy, for a total of up to 30 minutes.
Description: Participants were assessed for the following adverse events:
  * Decreased oxygen saturation
  * Increased respiratory rate
  * Increased heart rate
  * Low blood pressure
  * Increased work of breathing
  * Worsening arterial blood gases (if available)
  * Inability to tolerate the mouthpiece
Arm/Group | GO2 PEEP MOUTHPIECE
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GO2 PEEP MOUTHPIECE (N=2)
Decrease in oxygen saturation after cessation of PEEP therapy (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04331366/Prot_SAP_000.pdf